CLINICAL TRIAL: NCT07266493
Title: A Single-arm, Open-label, Single-center Prospective Study of Neoadjuvant Envafolimab Combined With Albumin-bound Paclitaxel and Carboplatin for Resectable Locally Advanced Esophageal Squamous Cell Carcinoma
Brief Title: Efficacy and Safety of Neoadjuvant Envafolimab Combined With Albumin-bound Paclitaxel and Carboplatin for Resectable Locally Advanced Esophageal Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Ge Di, Ge Di., MD, Shanghai Zhongshan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2023-222R
Record Dates: First submitted 2025-11-25; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Esophageal Squamous Cell Carcinoma; Neoadjuvant Therapy
Keywords: Esophageal Squamous Cell Carcinoma; Neoadjuvant therapy; Chemotherapy; Immunotherapy
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Carboplatin; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Envafolimab+Chemotherapy Group（EC Group） (Experimental): Envafolimab: 150mg, subcutaneous injection, administered on days 1, 8, and 15, treated for 3 weeks, followed by a 1-week rest period; Albumin bound paclitaxel: administered on days 1, 8, and 15, 100 mg/m2, IV , treated for 3 weeks, followed by a 1-week rest period; Carboplatin: administered on days 1, AUC 5, treated for 3 weeks, followed by a 1-week rest period. All patients will receive treatment with Envafolimab combined with albumin bound paclitaxel and carboplatin for three weeks, followed by one week of rest and a 28 day treatment cycle, for a total of two cycles. Then, the tumor condition of the patients will be evaluated to determine whether surgical treatment is feasible.
  Interventions: Drug: Chemotherapy （Albumin bound paclitaxel and Carboplatin）

INTERVENTIONS:
Drug: Chemotherapy （Albumin bound paclitaxel and Carboplatin） — Albumin bound paclitaxel: administered on days 1, 8, and 15, 100 mg/m2, IV , treated for 3 weeks, followed by a 1-week rest period; Carboplatin: administered on days 1, AUC 5, treated for 3 weeks, followed by a 1-week rest period.
  Other Names: Albumin bound paclitaxel and Carboplatin

SUMMARY:
This single center, prospective, single arm clinical study aims to evaluate the clinical efficacy and safety of Envafolimab combined with albumin bound paclitaxel and carboplatin as neoadjuvant therapy for locally advanced esophageal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* The subjects voluntarily joined this study, were able to sign the informed consent form, and had good compliance;
* Age ≥ 18 years old (when signing the informed consent form);
* ECOG score 0-1 points;
* Diagnosed with operable esophageal squamous cell carcinoma through pathological diagnosis (pathological tissue/cytology) and imaging;
* The clinical TNM staging is T2-4aNxM0
* Patients assessed to require routine neoadjuvant therapy;
* Have not received immunotherapy, chemotherapy, targeted therapy, or radiotherapy in the past;
* Expected survival ≥ 12 weeks

Exclusion Criteria:

* The subjects have any active autoimmune diseases or a history of autoimmune diseases (such as but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, pituitary inflammation, vasculitis, nephritis, thyroid dysfunction (hyperthyroidism/hypothyroidism), and the use of drugs cannot maintain thyroid function within the normal range, or patients who have undergone thyroid surgery and require long-term replacement therapy with thyroid hormone and other drugs after surgery); Subjects with vitiligo or complete remission of childhood asthma who do not require any intervention in adulthood may be included; Asthma in which subjects require bronchodilators for medical intervention cannot be included
* The subject has previous or concurrent malignant tumors;
* Patients who have received systemic anti-tumor therapy in the past;
* Individuals who have undergone significant surgical treatment, open biopsy, or significant traumatic injury within 28 days prior to the start of treatment; Or there may be wounds or fractures that have not been cured for a long time;
* There is a risk of bleeding, coagulation dysfunction, or currently undergoing thrombolytic therapy; Or have experienced esophageal or gastric variceal rupture bleeding in the past 6 months;
* It is known that the subject has a history of allergies to large molecule protein preparations or drug ingredients used;
* Subjects with any severe and/or uncontrolled illnesses
* Ascites or pleural effusion with clinical symptoms cannot be controlled with medication and require therapeutic puncture or drainage;
* The subject is known to have a history of substance abuse, alcoholism, or drug use;
* The researchers believe that participants should be excluded from this study, for example, if the researchers determine that there are other factors that may cause the study to be terminated midway

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate | From enrollment to the end of treatment at 8 weeks

SECONDARY OUTCOMES:
R0 resection rate | From enrollment to the end of treatment at 10 weeks
Major pathological response rate | From enrollment to the end of treatment at 8 weeks
ORR | From enrollment to the end of Cycle 2 (each cycle is 28 days)
  Objective response rate
3y-RFS rate | From enrollment until the date of first documented recurrence or date of death from any cause, whichever came first, assessed up to 36 months
  3-year recurrence free survival rate
3y-OS rate | From enrollment until the date of death from any cause, assessed up to 36 months
  3-year Overall survival rate

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No